CLINICAL TRIAL: NCT03991000
Title: Investigator-initiated, Randomized, Double-blind, Controlled, Multi-center Trial of Intravenous Iron in Patients With Cardiovascular Disease and Concomitant Iron Deficiency
Brief Title: Iron in Patients With Cardiovascular Disease
Acronym: iCHF-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to poor recruitment largely due to the covid pandemic, no safety concerns.
Sponsor: Dr. med. Mahir Karakas (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Mahir Karakas, Coordinating Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: iCHF-2
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Anemia, Iron-deficiency; Acute Myocardial Infarction; Atrial Fibrillation; Systolic Heart Failure
Keywords: Iron deficiency; Atrial fibrillation; Acute myocardial infarction; Systolic heart failure; Anemia
MeSH Terms: conditions — Cardiovascular Diseases; Anemia, Iron-Deficiency; Atrial Fibrillation; Heart Failure, Systolic; Iron Deficiencies; Anemia | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous iron (Experimental): Intravenous iron administration in the form of ferric carboxymaltose will be carried out according to summary of product characteristics. Bolus administration (1000 mg) will be followed by an optional administration of 500-1000 mg within the first 4 weeks (up to a total of 2000 mg which is in-label) according to approved dosing rules, followed by administration of 500 mg ferric carboxymaltose at months 4 and 8, except when haemoglobin is > 16.0 g/dL or ferritin is > 600 µg/L. To avoid unblinding in these patients a saline infusion will be administered.
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Administration of i.v. NaCl according to the dosing rules for intravenous iron.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous iron
  Arms: Intravenous iron
Drug: Saline — Saline application according to dosing rules of iron.
  Arms: Placebo

SUMMARY:
It is now recognized that iron deficiency in cardiovascular disease contributes to impaired clinical outcome.

DETAILED DESCRIPTION:
The clinical trial is designed as a prospective, multi-centre, double-blind, randomised, controlled, interventional trial to investigate whether a therapy with i.v. iron (iron carboxymaltose) compared to saline can improve functional status across a subset of cardiovascular disease -namely acute myocardial infarction, atrial fibrillation, and heart failure with reduced ejection fraction.

Iron administration will be carried out according to summary of product characteristics. Bolus administration (1000 mg) will be followed by an optional administration of 500-1000 mg within the first 4 weeks (up to a total of 2000 mg which is in-label) according to approved dosing rules, followed by administration of 500 mg iron carboxymaltose (over 15 minutes), except when haemoglobin is > 16.0 g/dL or ferritin is > 600 µg/L.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A (acute myocardial infarction): Acute Myocardial Infarction within 10 days (randomization/ first iron supplementation/ MRI must be performed within 10 days after AMI), without prior heart failure (defined as any known previous report of LVEF ≤ 45%) Cohort B (atrial fibrillation): Paroxysmal Atrial fibrillation or persistent AF Cohort C (heart failure): Left-ventricular ejection fraction ≤ 45 % (documented within the last 12 months prior to screening), all NYHA classes allowed
2. Confirmed presence of iron deficiency (ferritin < 100 ng/mL or ferritin 100 - 299 ng/mL with transferrin saturation < 20 %)
3. Haemoglobin ≤ 15.5 g/dL
4. Written informed consent

Exclusion Criteria:

1. Evidence of iron overload or disturbances in the utilisation of iron
2. History of severe asthma, eczema or other atopic allergy
3. History of immune or inflammatory conditions (e.g. systemic lupus erythematosus, rheumatoid arthritis)
4. Use of renal replacement therapy
5. Treatment with an erythropoietin stimulating agent (ESA), any i.v. iron and/or a blood transfusion in the previous 4 weeks prior to randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Cohort A: Left-ventricular ejection fraction | 16 weeks
  Change from baseline to week 16 in left-ventricular ejection fraction as determined by cardiac-MRI
Cohort B: Burden of atrial fibrillation | 12 months
  Delta between treatment groups in burden of atrial fibrillation from day 90 to 365 as assessed by a routinely implanted event recorder.
Cohort C: Left-ventricular ejection fraction | 16 weeks
  Change from baseline to week 16 in left-ventricular ejection fraction as determined by cardiac-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, MBA, Principal Investigator — University Heart Center Hamburg
Locations (3):
- Germany (3):
  - University of Berlin, Campus Benjamin-Franklin, Berlin
  - University Heart Center Hamburg, Hamburg
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No